CLINICAL TRIAL: NCT03993925
Title: Screening, Enhancement of Access to Care and Prioritization of Treatment for Chronic Hepatitis C Infection in High-risk Populations in Hong Kong
Brief Title: Enhancing Access to Care for Chronic Hepatitis C Infected Populations in Hong Kong
Status: Active, not recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Yuen Man Fung, Chair Professor of Gastroenterology and Hepatology, The University of Hong Kong
Other Study IDs: IN-HK-987-5354
Record Dates: First submitted 2019-06-18; First posted 2019-06-21 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Chronic Hepatitis C; Intravenous Drug Usage
Keywords: chronic hepatitis C; people who inject drugs; access to care; prison inmates
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Clotted blood will be stored for HCV RNA quantification and genotyping
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the current era of highly effective direct acting antiviral (DAA) therapy, the remaining obstacles to elimination of chronic HCV infection are identification of the high-risk groups, linkage to continued care and prevention of re-infection. It is estimated that 70-80% of patients with chronic HCV are unaware of their infection. Besides, public health education is limited and most patients are not aware that the current standard-of-care is highly effective, well tolerated and no longer require weekly subcutaneous injections. From a survey in Hong Kong in 2014, among 234 newly diagnosed HCV patients, only 20% agreed to undergo treatment. There is no universal screening programme for chronic hepatitis C infection in Hong Kong. and known high-risk patients include people who inject drugs (PWID), persons with certain medical conditions including those on hemodialysis, HIV infected, those with prior transfusion or organ transplantation. In this study, the investigators plan to reach out to PWIDs, people with substance abuse or prison inmates to provide rapid point-of-care screening for chronic hepatitis C infection, and to provide linkage to care for those diagnosed with chronic hepatitis C.

DETAILED DESCRIPTION:
Existing data on HCV sero-prevalence in these patients in Hong Kong is however fragmented especially in non-hospitalized persons. From the year 2014 surveillance report prepared by Department of Health (DH), anti-HCV prevalence rate among PWID under DH's methadone clinics was 46.2%. Two major issues remain in view of the high seroprevalence rate in this subgroup. Firstly, HCV RNA positivity was not reported and it is unknown whether these patients are still chronically infected. Many of patients are not directed to subsequent confirmatory tests and if they are chronically infected, they need to be linked to care. Secondly, data does not exist for these high-risk populations in Hong Kong. These subjects belong to high-risk group of harbouring undiagnosed chronic HCV and thus should be tested and linked to care.

Traditionally, the first step in screening for HCV utilizes enzyme immunoassay for the antibody against HCV. Fortunately, newer rapid diagnostic tests (RDT) can be used as a tool to screen subjects by providing point-of-care diagnosis on site. For instance, the OraQuick® HCV test (OraSure Technologies, Inc) is FDA-approved and CLIA-waived, with more than 98% sensitivity and specificity for qualitative detection of anti-HCV antibody in finger stick or venepuncture whole blood. As the volume of blood required is much smaller, subjects only need a finger stick for testing and results will be available within 20-40min. Subjects having positive results from RDT will proceed with venepuncture for collection of whole blood which will be sent back to our laboratory for confirmatory testing of anti-HCV antibody and HCV RNA.

Upon confirmation of diagnosis, subjects should be linked to care for further management. Ideally, all patients with chronic HCV should be treated regardless of severity of liver disease unless liver decompensation has developed necessitating liver transplantation before treatment or limited lifespan is expected even with DAA treatment. An integrated linkage-to-care clinic for all patients with newly diagnosed chronic HCV. Patients will be assessed in a timely manner. A dedicated research nurse will provide counselling and education to the patients. The nurse will then arrange on-site liver stiffness measurement with Fibroscan®, as well as phlebotomy for liver function test assessment.

This is a prospective cohort study. The investigators will form an outreach team and conduct visits to the relevant premises. The investigators will perform rapid diagnostic test (RDT) in high-risk populations. The investigators plan to conduct site visits every 4 - 8 weeks. The consent and potential impact of this study will be explained to subjects, followed by obtaining consent and blood taking. Subjects will also be asked to fill in a questionnaire, including information on age, gender, place of birth, ethnic origin, chronic medical illness, prior viral hepatitis infection, history of receiving HCV treatment and risk factors for contracting HCV (e.g. prior transfusion, intravenous drug use, tooth extraction or gum surgery, skin tattooing). Subjects will then have finger stick, which will be used for RDT as a point-of-care HCV screening test. If the RDT result is positive, the subject will then proceed with formal venepuncture for whole blood, which will be tested for confirmatory anti-HCV and HCV RNA (HCV genotype will also be determined for HCV RNA positive samples) in our own laboratory. The investigators will actively contact subjects confirmed with the diagnosis of chronic HCV. The research nurse will contact them to attend the integrated linkage-to-care clinic for counselling, education and risk stratification. During the clinic visits, risk stratification according to the liver status will be done by 1) physical examinations to document the clinical liver status, 2) comprehensive blood investigations including liver function tests, platelet counts and clotting profiles and 3) Fibroscan® to assess the fibrosis status. For institutionalised subjects, the invesrigators will conduct additional site visits for prescription and verification of SVR.

ELIGIBILITY:
Inclusion Criteria:

* People who inject drugs (PWID) who are receiving substance abuse counselling or rehabilitation treatment programs in halfway house and rehabilitation centres run by Non-governmental organisations (NGOs) in Hong Kong
* Prison inmates
* People with substance abuse

Exclusion Criteria:

* Already on antiviral therapy for known HCV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who inject drugs (PWID): receiving substance abuse counselling or rehabilitation treatment programs in halfway house and rehabilitation centres run by Non-governmental organisations (NGOs) in Hong Kong.
  Prison inmates: currently institutionalised under the Correctional Services Department.
  People with substance abuse: previous history or currently active substance abuse
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2019-09-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of newly diagnosed HCV patients being linked to care | 24 months
  Newly diagnosed HCV patients will be linked to local hepatologists for further treatment

SECONDARY OUTCOMES:
Prevalence rate of HCV in various high risk populations in Hong Kong | 24 months
  Prevalence rate of chronic hepatitis C infection in people who inject drugs/ prison inmates/ people with substance abuse
Proportion of various genotypes of HCV in PWIDs | 24 months
  Proportion of participants with various genotypes of chronic hepatitis C infection among PWIDs in Hong Kong

CONTACTS AND LOCATIONS:
Overall Officials: Man-Fung Yuen, DSc, MD, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Man Fung Yuen, Hong Kong, Please Select One ..., Hong Kong

IPD SHARING:
Plan to Share IPD: No